CLINICAL TRIAL: NCT01503801
Title: Inhaled Nitric Oxide to Prevent and Treat Bronchopulmonary Dysplasia in Preterm Infants
Brief Title: Inhaled Nitric Oxide to Prevent and Treat Bronchopulmonary Dysplasia
Acronym: NO-BPD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Children's Hospital of Fudan University (Other); Children's Hospital of Hebei Province (Other); Shen-Zhen City Maternity and Child Healthcare Hospital (Other); Hunan Children's Hospital (Other Government); QuanZhou Women and Children's Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Xiamen Women's and Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Bo Sun, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FudanU
Record Dates: First submitted 2011-12-19; First posted 2012-01-04 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Disease
Keywords: Preterm neonates; Bronchopulmonary dysplasia; Chronic lung disease; Inhaled nitric oxide; Respiratory therapy
MeSH Terms: conditions — Lung Diseases; Bronchopulmonary Dysplasia | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inhaled nitric oxide (Experimental): The preterm infants in the experimental group inhaled nitric oxide
  Interventions: Drug: Nitric Oxide
- oxygen (Active Comparator): The preterm infants enrolled but subjected to routine respiratory support.
  Interventions: Device: respiratory support

INTERVENTIONS:
Drug: Nitric Oxide — The infants in experimental group will receive inhale nitric oxide initiated at 5 ppm for 24 h followed by 2 ppm for 6 days or until weaning off
  Other Names: Nitrogen Monoxide; Endothelium Derived Relaxing Factor (EDRF)
  Arms: inhaled nitric oxide
Device: respiratory support — Routine respiratory support.
  Other Names: Nasal CPAP; Conventional mechanical ventilation; High frequency Oscillatory ventilation
  Arms: oxygen

SUMMARY:
Inhaled nitric oxide in preterm babies with respiratory failure or ventilator dependence will:

1. decrease the incidence of Bronchopulmonary Dysplasia (BPD) or death
2. shorten the length of oxygen therapy and hospital stay ,reduce the cost of hospital stay without increasing adverse effect

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia remains a problem in neonatal intensive care unit (NICU) all over the world. This multicenter, non-randomized, unmasked clinical trial evaluate the efficacy of inhaled nitric oxide (iNO) in the treatment of the preterm infant with developing bronchopulmonary dysplasia.

Infants were followed until death or discharge to home. The trial will compare iNO therapy to conventional management strategies (including treatment with nasal continuous positive airway pressure (CPAP), surfactant and high frequency ventilation as adjuncts to iNO therapy) as the control.

During the initial dosing, iNO was started at 5 ppm and could be decreased to 1-2 ppm. The Infants would inhale NO until weaned. Infants will be monitored for signs of toxicity due to cumulated dosage of NO and its metabolites, such as methemoglobin, and nitrite and nitrate in blood and urine, and nitrogen dioxide in ventilator circuit to the patient.

ELIGIBILITY:
Inclusion Criteria:

* GA<=34w,less than 7 days of age,oxygenation index (OI) of more than 10 after being ventilated for more than 48 hours or surfactant therapy
* GA<=34w,between 7 to 30 days of age, requiring assisted ventilator or nasal continuous positive airway pressure for more than 2 days

Exclusion Criteria:

* lethal congenital anomalies or congenital heart disease (including an atrial septal defect larger than 1 cm and a ventricular septal defect larger than 2 mm)
* active pulmonary hemorrhage, unevaluated pneumothorax
* preexisting bilateral grade 3-4 intraventricular hemorrhage
* a platelet count <100*10^9/l
* an expected duration of ventilation of less than 48 hours

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Death or Bronchopulmonary Dysplasia | Before discharge or at 36 weeks post-conceptional age
  the incidence of death before discharge or BPD at 36 weeks post-conceptional age

SECONDARY OUTCOMES:
Intraventricular Hemorrhage Grade III and IV | At 36 weeks post-conceptional age
  the incidence of Intraventricular Hemorrhage Grade III and IV At 36 weeks post-conceptional age
Days on assisted ventilation | Before discharge
  Days on assisted ventilation before discharge
Length of oxygen therapy | Before discharge
  Length of oxygen therapy before discharge
Retinopathy of prematurity | Before discharge
  Retinopathy of prematurity before discharge
Cost of hospital and NICU stay | Before discharge
  Medical cost of hospital and NICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Bo Sun, Ph.D, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China